CLINICAL TRIAL: NCT05281380
Title: Vitamin Insufficiency After Surgery for Esophagogastric Neoplasms: a Prospective Intervention Study
Brief Title: VITAMin Insufficiency in Esophagogastric Neoplasms
Acronym: VITAMIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL78919.096.21
Record Dates: First submitted 2021-10-21; First posted 2022-03-16 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Esophageal Cancer; Gastric Cancer; Vitamin Disease; Quality of Life
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with vitamin supplement (Other): Intervention with vitamin supplement Multi-E and Multi-G
  Interventions: Dietary Supplement: GIKAVI

INTERVENTIONS:
Dietary Supplement: GIKAVI — Two tailormade supplements for patients; one for that underwent esophagectomy and one for (sub-)total gastrectomy.

SUMMARY:
Rationale: Esophageal cancer and gastric cancer are among the top ten most common cancers worldwide. Both diseases have major impact on the nutritional status of patients and their quality of life. Studies investigating post-operative nutritional status are limited and postoperative identification and treatment of micro- and macronutritional deficiencies are currently lacking in (inter-)national guidelines.

Objective: To identify and target vitamin deficiencies after surgery for esophagogastric neoplasms.

Study design: Single centre intervention study. Study population: Patients aged 18 years and older that underwent esophagectomy or (sub- )total gastrectomy for esophagogastric neoplasms.

Intervention (if applicable): Two tailormade supplements for patients; one for that underwent esophagectomy and one for (sub-)total gastrectomy.

Main study parameters/endpoints: Baseline micronutrient deficiency measurements and after 6, 12, 24 months supplementation,.

Secondary study parameters/ endpoints: Occurrence of exocrine pancreatic insufficiency (n,%), occurrence of diarrhoea (n,%), steatorrhea (n,%), bloating (n,%), time between surgery and start of supplementation (mean in months), quality of life experienced (questionnaires) at baseline and after 6, 12, 24 months supplementation.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In this study, no health-related risks are present for participants due to the administration of supplementation that is already used as in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

A potential subject who meets any of the following criteria will be included for participation in this study:

* Patients ≥18 years of age who underwent an esophagectomy or (sub)total gastrectomy for malignancy with no signs of postoperative recurrence of disease.
* Written voluntary informed consent (IC).

Exclusion Criteria:

-

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Patients that underwent a wedge resection of the stomach
* Malignant disease recurrence
* Metastases
* Patients that are not capable to take supplementation due to altered mental status or swallow difficulties
* No signed informed consent
* Patients who are receiving chemotherapy
* Patients with high vitamin status at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Micronutrient deficiency yes or no. | 2 years
  Micronutrient deficiency yes or no.

SECONDARY OUTCOMES:
The incidence of exocrine pancreatic insufficiency | 2 years
  Faecal elastase test
To measure quality of life post-operative | 2 years
  Validated quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Guy Vijgen, MD,PhD, Principal Investigator — Zuyderland MC
Locations (1):
- ZuyderlandMC, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Velden AL, Vermeer TA, Boerma EG, Belgers EH, Stoot JH, Leers MP, Sosef MN, Vijgen GH. Vitamin insufficiency after surgery for oesophagogastric neoplasms: a study protocol for a prospective intervention study. BMJ Open. 2023 Jul 4;13(7):e067981. doi: 10.1136/bmjopen-2022-067981. PMID 37407040